CLINICAL TRIAL: NCT02104492
Title: Clinical Research on the Effect of a 12-week Respiratory Muscles Training Program in Persons With Relapsing-remitting Multiple Sclerosis
Brief Title: Effects of a 12-week Respiratory Muscles Training Program in Persons With Relapsing- Remitting Multiple Sclerosis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Malaga (Other)
Responsible Party: Principal Investigator, Rocío Martín Valero, Ph D, University of Malaga
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: UMA_RMTP_2014/SM; Respiratory Sclerosis Multple (Other: RESM)
Record Dates: First submitted 2014-03-27; First posted 2014-04-04 (Estimated); Last update posted 2014-04-04 (Estimated); Status verified 2014-04

CONDITIONS: Relapsing-remitting Multiple Sclerosis
Keywords: multiple sclerosis; respiratory muscle strength; maximal inspiratory pressure (MIP); maximal expiratory pressure (MEP); respiratory muscle endurance; quality of life; qualitative research
MeSH Terms: conditions — Multiple Sclerosis, Relapsing-Remitting; Multiple Sclerosis | interventions — Control Groups

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Intervention group (Experimental): a 12-week respiratory muscles training program (RMTP) with ORYGEN Dual® device and peripheric resistive muscle training program
  Interventions: Other: a 12-week Respiratory Muscles Training Program (RMTP)
- Control Group (Active Comparator): Peripheric resistive muscle training program and Health Education Program.
  Interventions: Other: Active Comparator

INTERVENTIONS:
Other: a 12-week Respiratory Muscles Training Program (RMTP) — Every session will be lasted 50 minutes and performed under supervision of a physiotherapist. It will be comprised of 30 minutes of progressive aerobic training program followed by peripheric resistive muscle training program which will be supplemented by a 12-week Respiratory Muscles Training Program (RMTP) with ORYGEN Dual® device for 20 minutes. Patients will be instructed to maintain adequate inspiration and expiration while using the Origen-Dual® valve at a rate of 15-20 breaths/minute. Participants will be performed five sets of 10 repetitions followed by 1-2 minutes of unloaded recovery breathing off the device, once a day, 2 days per week, for 12 weeks. The respiratory muscles training will be begun at 30% of MIP achieved at baseline and increased by 5% each week to reach 60% of the baseline assessment MIP.
  Other Names: Intervention Group
  Arms: Intervention group
Other: Active Comparator — Every session will be comprised of 30 minutes of progressive aerobic training program followed by peripheric resistive muscle training program and Health Education Program.
  Other Names: Control Group
  Arms: Control Group

SUMMARY:
Multiple sclerosis (MS) is the most common inflammatory demyelinating chronic disease of the central nervous system and the second leading cause of disability in young adults. Motor deficits also involve respiratory muscles. This involvement is present from early stages of disease and is frequently dismissed by professionals until advanced stages of disease. The effect of a training program of respiratory muscles is not sufficiently studied. The aim of this research is to assess the clinical and functional response of a 12-week respiratory muscles training program (RMTP) for persons with relapsing-remitting multiple sclerosis (RRMS).

This study is consisted with two sub research:

Firstly, a single-blind randomized clinical trial will be carried out in 40 persons with RRMS. Participants either will be received (n = 20) peripheric resistive muscle training program which will be supplemented by a 12-week Respiratory Muscles Training Program (RMTP) with ORYGEN Dual® device for 50 minutes, twice a week during three months or (n = 20) they will be received peripheric resistive muscle training program and health education program. Main outcomes will be strength of the respiratory muscles assessed by maximal inspiratory and expiratory pressure measurements (MIP and MEP). The secondary outcomes will be assessed the quality of life (MSQOL-54), walking speed (T25-FW, MSWS-12 and Hauser ambulatory index), fatigue (MFIS), endurance of the respiratory muscles (10RM) manoeuvre and peripherical muscle strength (Multiple-Sit-to-Stand Test and handgrip strength).

Secondly, the qualitative research where researchers will interview participants about their interest in carrying out the intervention (difficulties and advantages) and identify themes of interest about changes in quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Males and females older 18 years of age with diagnosis relapsing-remitting multiple sclerosis according to revised McDonald Criteria 2005.
* Have mild or moderate impairment of gait according to Hauser ambulatory index. The score 1 and 5 will be included (both values inclusive).
* Subjects who have read, understood, signed and dated the informed consent form.

Exclusion Criteria:

* Disability caused by other diseases
* Clinically relevant cognitive or linguistic disorders which are unable to fill in the questionnaires by him/herself
* Subjects used medication with corticosteroids within the last month (or 30 days) prior to study day 1.
* Have a recent outbreak (last month) not stabilized prior to inclusion in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2014-03; Primary Completion 2015-03 (Estimated); Study Completion 2015-03 (Estimated)

PRIMARY OUTCOMES:
Maximal inspiratory pressures (MIP) and maximal expiratory pressures (MEP) | Baseline and 12 weeks
  Change in respiratory muscle function strength with transducer measuring maximal inspiratory (MIP) and expiratory pressures (MEP)

SECONDARY OUTCOMES:
Pulmonary function test | Baseline and 12 weeks
  Pulmonary function test will be performed using spirometer "DATOSPIR 120" according to the Guidelines of American Thoracic Society and the European Respiratory Society.
Handgrip strength | Baseline and 12 weeks
  Handgrip strength will be determined using hydraulic hand dynamometer "JAMAR"
Multiple-Sit-to-Stand Test (MSTS) | Baseline and 12 weeks
  Lower limb strength using the Multiple-Sit-to-Stand Test (MSTS)
The 12 item MS Walking Scale (MSWS-12) | Baseline and 12 weeks
  Walking Capacity using the 12 item MS Walking Scale (MSWS-12)
Timed 25 foot walk (T25FW) | Baseline and 12 weeks
  Exercise Capacity using the Shorter timed walking tests with Timed 25 foot walk (T25FW)
Gait analysis | Baseline and 12 weeks
  Gait analysis (the Hauser ambulatory index) with which will be assessed the time and effort used by the patient to walk 25 feet (8 meters)
The 54 items Specific Questionnaire Quality of Life Multiple Sclerosis (MSQOL-54) | Baseline and 12 week
  Change in quality of life using the 54 items Specific Questionnaire Quality of Life Multiple Sclerosis (MSQOL-54)
10 Maximum Resistance (10RM) | Baseline, 4 weeks, 8 weeks, 12 weeks.
  Change in endurance of the respiratory muscles with the 10RM manoeuvre
Perceptions Measures | 12 weeks
  Post interview with participants to qualitatively identify themes of interest and quality of life effects After that the respiratory muscles training program, researchers will interview participants about their interest in carrying out the intervention (difficulties and advantages) and changes in quality of life

CONTACTS AND LOCATIONS:
Locations (1):
- University of Málaga, Málaga, Málaga, Spain